CLINICAL TRIAL: NCT04336449
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Single-ascending-dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Eptinezumab in Healthy Japanese Subjects
Brief Title: Eptinezumab in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18899A
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 100 mg eptinezumab (Experimental)
  Interventions: Drug: Eptinezumab
- Cohort 2 300 mg eptinezumab (Experimental)
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Eptinezumab - single intravenous infusion
  Arms: Cohort 1 100 mg eptinezumab; Cohort 2 300 mg eptinezumab
Drug: Placebo — Placebo - single intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate how eptinezumab enters, moves through and exits the body. Safety and tolerability will also be investigated.

DETAILED DESCRIPTION:
The study will consist of 18 healthy Japanese subjects, divided into two single dose cohorts with 9 subjects in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese subjects with a BMI of ≥ 18.5 and ≤ 25 kg/m2

Other in- and exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Cmax eptinezumab | From dosing to week 12
  maximal observed plasma concentration
AUC(0-t) eptinezumab | From dosing to week 12
  area under the plasma concentration-time curve from zero to time t
AUC(0-inf) eptinezumab | From dosing to week 12
  area under the plasma concentration-time curve from zero to infinity
Systemic Clearance of eptinezumab | From dosing to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- P-One Clinic, Tokyo, Japan